CLINICAL TRIAL: NCT04084990
Title: Sleep Apnea and Fetal Growth Restriction
Acronym: SAFER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to insufficient recruitment.
Sponsor: Washington University School of Medicine (Other)
Collaborators: ResMed Foundation (Other); Hebrew University Hadassah Medical School (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Alexander M. Hincker, Assistant Professor, Department of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201908162
Record Dates: First submitted 2019-09-07; First posted 2019-09-11 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Obstructive Sleep Apnea; Fetal Growth Restriction; Pregnancy Related
Keywords: aPAP; OSA; FGR
MeSH Terms: conditions — Sleep Apnea, Obstructive; Fetal Growth Retardation

STUDY DESIGN:
Intervention Model Description: Prospective, parallel group, investigator-blinded, randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- aPAP (Experimental): Nightly use of aPAP when sleeping through the date of delivery
  Interventions: Device: S9 VPAP Adapt
- No aPAP (No Intervention): No use of aPAP (standard of care)

INTERVENTIONS:
Device: S9 VPAP Adapt — Auto-titrated positive airway pressure
  Arms: aPAP

SUMMARY:
This study aims to evaluate the association between obstructive sleep apnea (OSA) and fetal growth restriction (FGR) and to assess the role of auto-titrated positive airway pressure (aPAP) as antenatal therapy in these patients. Pregnant patients with diagnosed FGR will be screened for OSA first by screening questionnaire and then by home sleep monitor. Of those patients diagnosed with OSA, half will be assigned to use aPAP each night when sleeping and half will not (standard care).

DETAILED DESCRIPTION:
Fetal growth restriction (FGR) affects 5-10% of pregnancies and is one of the leading causes of perinatal morbidity and mortality.

Obstructive sleep apnea (OSA) is a common disorder in which a person's breathing pauses or becomes shallow during sleep. These periods of low oxygen lead stress and inflammation which that may be harmful to both the mother and her fetus. OSA in pregnancy has been associated with poor maternal-fetal outcomes, including low birth weight, preterm delivery, FGR, gestational hypertension/preeclampsia, gestational diabetes and higher rates of neonatal ICU admission.

Auto-titrated positive airway pressure (aPAP) is a machine that gently delivers pressurized air via a mask to keep a patient's airways free of obstruction during sleep. It is currently unclear whether treatment of OSA during pregnancy in women with known FGR can improve fetal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 50
* Fetal growth restriction (defined as fetal weight <10th percentile based on at least one routine 2nd trimester ultrasound without a subsequent increase to >15th percentile on any ultrasounds prior to enrollment)
* Lower limit of gestational age at enrollment 22+0 weeks.
* Upper limit of gestational age at enrollment: adequate time to complete Stages 1 and 2 and if appropriate to be randomized and receive intervention by no later than 32+0 weeks.
* The absence of 2 minor or 1 major markers of aneuploidy.

Exclusion Criteria:

* Other known cause of fetal growth restriction (including congenital anomalies, intrauterine infection, or multiple gestation)
* Reversed end-diastolic flow in the umbilical artery
* Preexisting diagnosis of OSA being treated with aPAP
* Chronic pulmonary disease (cystic fibrosis, moderate persistent asthma)
* Hemoglobinopathies (sickle cell anemia, thalassemia)
* Maternal craniofacial anomalies
* Premature rupture of membranes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hincker, MD, Principal Investigator — Washington University in Saint Louis
Locations (3):
- United States (2):
  - Washington University in St. Louis, St Louis, Missouri
  - Rochester University Medical Center, Rochester, New York
- Hadassah Hebrew University, West Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Nardozza LM, Caetano AC, Zamarian AC, Mazzola JB, Silva CP, Marcal VM, Lobo TF, Peixoto AB, Araujo Junior E. Fetal growth restriction: current knowledge. Arch Gynecol Obstet. 2017 May;295(5):1061-1077. doi: 10.1007/s00404-017-4341-9. Epub 2017 Mar 11. PMID 28285426
- [Background] Lavie L. Oxidative stress in obstructive sleep apnea and intermittent hypoxia--revisited--the bad ugly and good: implications to the heart and brain. Sleep Med Rev. 2015 Apr;20:27-45. doi: 10.1016/j.smrv.2014.07.003. Epub 2014 Jul 24. PMID 25155182
- [Derived] Hincker A, Nadler J, Karan S, Carter E, Porat S, Warner B, Ju YS, Ben Abdallah A, Wilson E, Lockhart EM, Ginosar Y. Sleep Apnea and Fetal Growth Restriction (SAFER) study: protocol for a pragmatic randomised clinical trial of positive airway pressure as an antenatal therapy for fetal growth restriction in maternal obstructive sleep apnoea. BMJ Open. 2021 Jun 29;11(6):e049120. doi: 10.1136/bmjopen-2021-049120. PMID 34187829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has been terminated due to low enrollment after only 3 participants were randomized. Results will not be analyzed owing to the small number of participants to be randomized to receive aPAP (the intervention) or no aPAP (standard of care treatment).
Pre-assignment Details: 32 participants provided informed consent to participate. They underwent an obstructive sleep apnea (OSA) risk assessment questionnaire. Those screening as high risk for OSA underwent home sleep apnea testing (HSAT). Those screening as positive on the HSAT, which was defined as an apnea hypopnea index (AHI) >= 10 OR an AHI >= 5 with oxygen desaturation index >= 5, were randomized to receive aPAP or not. Of the 32 participants, only 3 met criteria for enrollment in the randomization phase.
Period: Overall Study
Arm/Group | aPAP | No aPAP
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | aPAP | No aPAP | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 32.8 [32.2 to 33.4] | 29.8 [29.8 to 29.8] | 31.8 [29.8 to 33.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Birth Weight
Description: Weight of child at time of birth
Time Frame: 1 day
Population: Of two mothers randomized to aPAP therapy, one required pre-term induction of labor for maternal safety for preeclampsia with severe features. This fetus experienced in-utero fetal demise, so birth weight was not obtained.
Measure: Mean (Full Range); unit: grams
Arm/Group | aPAP | No aPAP
Number analyzed (Participants) | 1 | 1
grams | 2320 [2320 to 2320] | 570 [570 to 570]

2. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age at delivery
Time Frame: 1 day
Measure: Mean (Full Range); unit: weeks (estimated gestational age)
Arm/Group | aPAP | No aPAP
Number analyzed (Participants) | 2 | 1
weeks (estimated gestational age) | 31.4 [25.7 to 37.1] | 25.7 [25.7 to 25.7]

ADVERSE EVENTS:
Time Frame: Approximately 9.5 months
Arm/Group | aPAP | No aPAP
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT04084990/Prot_SAP_003.pdf
  • Informed Consent Form (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT04084990/ICF_001.pdf